CLINICAL TRIAL: NCT06876545
Title: Identification of Vitamin C Deficiency in Hospitalized Adults Through a Systematic Approach Vs. Traditional Medical Judgment: a Before-and-After Observational Study
Brief Title: "Vitamin C Deficiency in Hospitalized Adults: Systematic Screening Vs. Traditional Judgment - a Before-and-After Observational Study"
Status: Not yet recruiting | Type: Observational
Sponsor: Internist.Ro (Other)
Collaborators: Centre Hospital Regional Universitaire de Limoges (Other)
Responsible Party: Principal Investigator, Purcarea Adrian, MD, PhD, Internist.Ro
Other Study IDs: A001
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Scurvy
Keywords: Scurvy, vitamin C defficiency, hospitalized
MeSH Terms: conditions — Scurvy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Historical control group: Control Group (Historical Cohort):
  Patients who underwent Vitamin C testing based on traditional clinical judgment, meaning testing was performed "as needed" at the discretion of the treating physician.
  No standardized criteria were applied for selecting patients for Vitamin C testing.
  Data will be collected from medical records retrospectively (prior to the introduction of a systematic screening approach).
- Prospective Cohort: Active Group (Systematic Screening Cohort):
  Patients who underwent Vitamin C testing based on a predefined, rigorous suspicion framework (SFI - Scurvy Suspected upon Hemorrhagic Risk).
  Testing was systematically performed in patients with predefined hemorrhagic risk factors, including:
  Hematuria (macroscopic or detected via dipstick/microscopy). Ecchymoses (bruising). Petechiae. Epistaxis. Gastrointestinal bleeding (melena, hematemesis, positive fecal occult blood test).
  Cerebral hemorrhage. The selection for testing was systematic and protocol-driven, ensuring a more structured and standardized approach.
  Interventions: Diagnostic Test: systematical screening of at risk patients based on predefined hemorrhagic criteria

INTERVENTIONS:
Diagnostic Test: systematical screening of at risk patients based on predefined hemorrhagic criteria — Patients selected if condition present:
  Hematuria (blood in urine)
  Macroscopic hematuria (visible blood in urine) Hematuria detected by urine dipstick or microscopic analysis Ecchymoses (bruising)
  Epistaxis (nosebleeds)
  Petechiae (small pinpoint hemorrhages on the skin)
  Gastrointestinal bleeding
  Upper GI bleeding: Hematemesis (vomiting blood) Lower GI bleeding: Melena (black tarry stools) Positive fecal occult blood test (FOBT) Cerebral hemorrhage (brain bleeding)
  Groups: Prospective Cohort

SUMMARY:
Brief Summary of the Study The goal of this observational study is to assess the incidence of vitamin C deficiency among hospitalized adults presenting with hemorrhagic signs. The study will also evaluate the effectiveness of a standardized screening protocol compared to traditional clinical judgment.

The main questions it aims to answer are:

What is the incidence of vitamin C deficiency in hospitalized patients with hemorrhagic symptoms? Is a standardized screening protocol more effective than traditional clinical judgment in identifying vitamin C deficiency? Is vitamin C deficiency associated with anemia, other micronutrient deficiencies (folate, B12, albumin, iron), or infectious conditions? Does vitamin C deficiency impact hospital length of stay? Researchers will compare a systematic screening approach based on predefined hemorrhagic criteria (e.g., hematuria, ecchymosis, epistaxis, petechiae, gastrointestinal bleeding, or intracranial hemorrhage) to the traditional physician-judgment approach to determine its effectiveness in identifying vitamin C deficiency.

Study Design

Participants will:

Be hospitalized adults (≥18 years old) presenting with documented micro- or macroscopic hemorrhagic signs.

Undergo vitamin C level assessment either as part of the standardized screening protocol (prospective arm) or based on physician judgment (retrospective control group).

Have additional clinical and laboratory data collected, including hemoglobin levels, platelet count, iron status, vitamin B9/B12 levels, and other relevant parameters.

This non-interventional study will not modify the standard of care but will systematically assess the prevalence of vitamin C deficiency in at-risk patients and evaluate the utility of a structured screening protocol.

DETAILED DESCRIPTION:
Study Design and Methodology

Study Type:

Observational (before-after study design)

Retrospective for the control group (patients with historical vitamin C measurements) and for exposure group (patients systematically screened based on predefined hemorrhagic criteria)

Study Population:

Inclusion Criteria:

Adults (age ≥18 years) admitted to the hospital

Presence of micro- or macroscopic hemorrhagic symptoms

Undergoing vitamin C level assessment (either systematic or based on physician discretion)

Exclusion Criteria:

Refusal to participate

Prior vitamin C supplementation within one month before the study period

Study Groups:

Control Group (Retrospective):

Patients with documented hemorrhagic symptoms for whom vitamin C levels were measured based on physician judgment (prior to implementation of systematic screening criteria).

Exposure Group (Prospective):

Patients identified through a systematic screening protocol incorporating predefined hemorrhagic criteria.

Primary Outcome:

Incidence of vitamin C deficiency (defined as serum ascorbic acid levels below laboratory reference ranges) in patients with hemorrhagic symptoms.

Secondary Outcomes:

Diagnostic efficiency of the systematic screening approach versus traditional physician-led assessment.

Association between vitamin C deficiency and anemia (hemoglobin levels, mean corpuscular volume, ferritin, reticulocyte count, transferrin saturation).

Association with other micronutrient deficiencies (folate, B12, albumin, and iron status).

Presence of concurrent infections in vitamin C-deficient patients.

Impact on hospital length of stay in vitamin C-deficient patients versus non-deficient patients.

Data Collection and Registry Procedures

Quality Assurance Plan:

Data validation and registry procedures include automated and manual data checks for completeness and consistency.

On-site data audits will be conducted to ensure compliance with study protocols.

Standardized case report forms (CRFs) will be used for data collection.

Data Verification and Source Validation:

Data consistency checks will compare registry entries with patient medical records.

Laboratory values will be cross-validated against hospital electronic records.

External source verification will be conducted for select cases to assess data accuracy.

Standard Operating Procedures (SOPs):

Patient Recruitment: Patients meeting inclusion criteria will be identified through hospital electronic records and physician referrals.

Data Collection:

Baseline assessment will include demographic details, medical history, and medication use (e.g., anticoagulants, nutritional supplements).

Clinical evaluation will include hemorrhagic symptoms (ecchymosis, petechiae, gastrointestinal bleeding, hematuria, epistaxis).

Laboratory assessments will include vitamin C levels, hemoglobin, ferritin, folate, B12, albumin, and markers of infection.

Data Management:

De-identified patient data will be stored in a secure, access-controlled database.

Routine data audits will ensure quality and completeness.

Statistical Analysis:

Data will be analyzed per predefined statistical models to assess prevalence and associations.

Sample Size Assessment:

Estimated 42 patients per group based on prevalence estimates of 20% vitamin C deficiency in hospitalized patients with hemorrhagic symptoms.

Sample size determination accounts for a power of 80% and alpha of 0.05.

Bayesian inference will be applied if sample size calculations require adjustments based on interim analyses.

Plan for Handling Missing Data:

Imputation methods (multiple imputations) will be used for missing laboratory values.

Sensitivity analyses will assess the impact of missing data on study conclusions.

Statistical Analysis Plan:

Descriptive Statistics:

Mean, median, standard deviation for continuous variables.

Frequency distribution for categorical variables.

Comparative Analyses:

Student's t-test or Mann-Whitney U test for continuous variables.

Chi-square or Fisher's exact test for categorical variables.

Multivariable Regression Models:

Adjustments for confounders (age, comorbidities, nutritional status, anticoagulant use).

Logistic regression for risk factor analysis of vitamin C deficiency.

Cox proportional hazards model for hospital length of stay impact analysis.

Sensitivity Analyses:

Assess variations in vitamin C deficiency prevalence.

Evaluate changes in detection efficiency of systematic screening protocol.

Ethical Considerations

The study is non-interventional and does not alter clinical care.

Patient confidentiality will be ensured through anonymized data collection and secure storage.

Informed consent will be obtained for prospective participants.

The study has received ethical approval from the Centre Hospitalier de Guéret Ethics Committee.

Data Dissemination Plan

Results will be published in peer-reviewed medical journals.

Findings will be shared with hospital medical teams to optimize patient care.

A summary report will be provided to participants upon study completion.

Conclusion

This study will provide critical insights into the prevalence of vitamin C deficiency in hospitalized patients with hemorrhagic symptoms. By evaluating a structured screening approach, this research aims to improve early detection and clinical awareness of vitamin C deficiency, potentially informing future guidelines for at-risk populations.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized adult patients (≥18 years old) who had Vitamin C testing performed during their hospital stay.

Documented hemorrhagic manifestations in medical records, including at least one of the following:

Hematuria (macroscopic or detected via urine dipstick/microscopy). Ecchymoses (bruising). Petechiae. Epistaxis (nosebleeds). Gastrointestinal bleeding (melena, hematemesis, or positive fecal occult blood test).

Cerebral hemorrhage. Medical records available with sufficient clinical and laboratory data to assess eligibility and study variables.

Patients from two distinct periods:

Historical Control Group: Patients tested for Vitamin C "as needed" based on traditional medical judgment.

Active Group: Patients tested systematically according to Scurvy Suspicion upon Hemorrhagic Risk (SFI) criteria after protocol implementation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received Vitamin C supplementation within the month prior to testing.
  Incomplete or missing medical records regarding hemorrhagic manifestations or Vitamin C test results.
  Hemorrhagic events clearly attributable to anticoagulant or antiplatelet overdose, without other potential contributing factors.
  Blood samples processed more than 2 hours after collection, making Vitamin C levels unreliable.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of the study is the existence of Vitamin C deficiency in hospitalized patients presenting with hemorrhagic signs. | The total study duration is expected to be around 4 months (3 months retrospective + 1 month prospective), but data collection may continue if necessary to reach the required sample size.
  Definition of the Primary Outcome:
  Vitamin C deficiency will be determined based on serum ascorbic acid levels measured through blood sampling.
  A deficient status is defined as a serum ascorbic acid concentration below the reference values established by the central laboratory (Cerba, Paris, France).
  Only samples processed within 2 hours of collection will be considered valid due to the instability of ascorbic acid.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Purcarea MD, Study Director — Transylvania Univeristy, Faculty of Medicine, Brasov, Romania; Silvia Sovaila MD, Principal Investigator — Transylvania Univeristy, Faculty of Medicine, Brasov, Romania; Remy Bouquet MD, Principal Investigator — Gueret Hospital, Creuse, France
Locations (1):
- Gueret Hospital, Guéret, Creuse, France

IPD SHARING:
Plan to Share IPD: Yes
If justified and after accord from the local Ethics Committee
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 10years after study start
Access Criteria: If justified by formal request or predefined protocol and after accord from the local Ethics Committee